CLINICAL TRIAL: NCT03482141
Title: Clinical Utility of Prenatal Whole Exome Sequencing
Acronym: PWES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-22420
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Structural Anomalies; Cardiac Anomalies; Central Nervous System Anomalies; Thorax Anomalies; Genito-urinary Anomalies; Gastrointestinal Anomalies; Skeletal Anomalies; Multiple Anomalies
MeSH Terms: conditions — Heart Defects, Congenital; Abnormalities, Multiple | interventions — Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Whole Exome Sequencing (Other): Whole exome sequencing (WES) will take place for prenatal patients (pregnancies with fetal structural defects). All patients will get exome sequencing and will follow the same procedures.
  Interventions: Device: Whole Exome Sequencing (WES)

INTERVENTIONS:
Device: Whole Exome Sequencing (WES) — The Investigators will enroll pregnant women with fetal anomalies detected by ultrasound. Patients will be approached by a maternal-fetal specialist, who has counseled the patient regarding the fetal anomaly that has been detected. Written informed consent will be obtained by the study prenatal genetic counselor. Many patients will have undergone prenatal diagnostic testing in an outside laboratory; in such cases, cells or extracted DNA from the original fetal sample will be used for the purpose of this study. The consent process for prenatal WES will include pre-test counseling and the option of choosing whether or not to receive uncertain results and secondary findings. After conducting whole exome sequencing, the findings will be shared with the parent(s). Routine medical care will be provided to patients. The research will study the effectiveness of sequencing as a tool for providing genetic information to parents when a prenatal study reveals a fetus with a structural anomaly.

SUMMARY:
The investigator aims to examine the clinical utility of WES, including assessment of a variety of health-related and reproductive outcomes in undiagnosed prenatal cases.

DETAILED DESCRIPTION:
Next-generation sequencing (NGS) is changing the paradigm of clinical genetic testing. Unlike highly focused single-gene tests, NGS allows one to examine gene panels, the exome, and the whole genome. With the broad array of molecular tests now available, ordering physicians face the conundrum of selecting the best diagnostic tool for patients with suspected genetic conditions. Single-gene testing is often most appropriate for conditions with distinctive clinical features and minimal locus heterogeneity. NGS-based gene panel testing, which can be complemented with chromosomal microarray analysis (CMA) and other ancillary methods, provides a comprehensive and feasible approach for well documented but genetically heterogeneous disorders. Whole exome sequencing (WES) and whole genome sequencing (WGS) have the advantage of enabling parallel interrogation of most of the genes in the human genome. To some, WES is preferable to previously used methods due to higher diagnostic yield, shorter time to diagnosis, and improved cost-efficiency.

The ability to survey the exome opens up both new opportunities and new challenges. For example, all coding regions of known genes must be analyzed when applying WES to undiagnosed cases with unclear inheritance patterns. Current limitations on variant interpretation capabilities and clinical validity raise questions about the clinical utility of WES as either a stand-alone or a first-choice diagnostic test. Additional challenges include pre- and post-test counseling with appropriate and robust informed consent, bioinformatics analysis setup and validation, variant interpretation and classification, the need for policies and protocols concerning the discovery and reporting of secondary findings unrelated to the presenting indication, a requirement for validation of WES results, assurance of conformation to quality control standards, data storage and accessibility, and reimbursement issues.

Current clinical standards recommend offering chromosomal microarray (CMA) in the prenatal setting when fetal structural anomalies are detected via prenatal ultrasound. In these cases, clinically relevant copy number variants have been reported in 6.0-9.1% of fetuses with a normal karyotype. However, informed consent processes for prenatal CMA are challenging-particularly in cases with ultrasound anomalies, as parents are absorbing challenging news and under considerable stress. Women have reported being "blindsided" by positive CMA results, or feeling that these results were "toxic information"-information they wished they did not have, particularly in cases of uncertain genetic information or uninterpretable variants. Nonetheless, in that same study women who were referred for CMA because of ultrasound anomalies reported less frequent negative reactions, since they already anticipated abnormal results.

Introducing WES into prenatal clinical care of underrepresented populations raises additional issues and considerations of payment coverage, access, and standards of care. Beyond the sheer complexity of the test and its results, clinicians and health systems must address numerous considerations, including: private and public insurance coverage; language and culture differences and their implications for genetic counseling and clinician-patient relationships; ability to access follow-up testing and clinical care; ability to access appropriate treatment and services; and particularly in the prenatal setting, local, state, and national abortion laws and decision-making about pregnancy termination. These issues and others will affect not only patients' decision-making regarding WES, but also their post-test needs for patient follow up, counseling and support. The importance of systematically assessing the clinical utility of NGS is critical for determining in which clinical and health care contexts WES will be useful and for commencing research on these considerations.

The investigator aims to examine the clinical utility of WES, including assessment of a variety of health-related and reproductive outcomes in undiagnosed prenatal cases.

ELIGIBILITY:
Inclusion Criteria:

* Women carrying a pregnancy with an ultrasound diagnosis of a major structural anomaly (or multiple anomalies) in a major organ system (cardiac, central nervous system, thorax, genito-urinary, gastrointestinal/ventral wall, skeletal and or multiple anomalies )
* Clinical concern for a potential underlying genetic condition
* Completed or plan to complete chorionic villus sampling or amniocentesis with chromosome analysis or microarray
* Available maternal sample

Exclusion Criteria:

* Prior WES performed for a clinical or research indication
* Lack of phenotypic indication of a likely underlying genetic etiology
* Mother unwilling or unable to provide a specimen

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 316 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Norton, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Muzny DM, Reid JG, Bainbridge MN, Willis A, Ward PA, Braxton A, Beuten J, Xia F, Niu Z, Hardison M, Person R, Bekheirnia MR, Leduc MS, Kirby A, Pham P, Scull J, Wang M, Ding Y, Plon SE, Lupski JR, Beaudet AL, Gibbs RA, Eng CM. Clinical whole-exome sequencing for the diagnosis of mendelian disorders. N Engl J Med. 2013 Oct 17;369(16):1502-11. doi: 10.1056/NEJMoa1306555. Epub 2013 Oct 2. PMID 24088041
- [Background] Norton ME, Rink BD. Changing indications for invasive testing in an era of improved screening. Semin Perinatol. 2016 Feb;40(1):56-66. doi: 10.1053/j.semperi.2015.11.008. Epub 2015 Dec 24. PMID 26725145
- [Background] Cowan RS. Aspects of the history of prenatal diagnosis. Fetal Diagn Ther. 1993 Apr;8(Suppl. 1):10-7. doi: 10.1159/000263869. PMID 11653011
- [Background] Chervenak FA, McCullough LB. Ethical issues in perinatal genetics. Semin Fetal Neonatal Med. 2011 Apr;16(2):70-3. doi: 10.1016/j.siny.2010.10.004. Epub 2010 Nov 3. PMID 21051301
- [Background] Donley G, Hull SC, Berkman BE. Prenatal whole genome sequencing: just because we can, should we? Hastings Cent Rep. 2012 Jul-Aug;42(4):28-40. doi: 10.1002/hast.50. Epub 2012 Jun 20. PMID 22777977
- [Derived] Rego S, Hoban H, Outram S, Zamora AN, Chen F, Sahin-Hodoglugil N, Anguiano B, Norstad M, Yip T, Lianoglou B, Sparks TN, Norton ME, Koenig BA, Slavotinek AM, Ackerman SL. Perspectives and preferences regarding genomic secondary findings in underrepresented prenatal and pediatric populations: A mixed-methods approach. Genet Med. 2022 Jun;24(6):1206-1216. doi: 10.1016/j.gim.2022.02.004. Epub 2022 Apr 8. PMID 35396980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited prenatal patients to this study and completed exome sequencing with 316 cases.
Pre-assignment Details: This is an exploratory study to define the diagnostic yield of exome sequencing in a prenatal population. All participants were offered the same test and received the same study procedures. There are no arms in this study.
Groups:
- Whole Exome Sequencing: Whole exome sequencing (WES) will take place for all enrolled patients.
  The Investigators will enroll pregnant women with fetal anomalies detected by ultrasound. Patients will be approached by a maternal-fetal specialist, who has counseled the patient regarding the fetal anomaly that has been detected. Written informed consent will be obtained by the study prenatal genetic counselor. Many patients will have undergone prenatal diagnostic testing in an outside laboratory; in such cases, cells or extracted DNA from the original fetal sample will be used for the purpose of this study. The consent process for prenatal WES will include pre-test counseling and the option of choosing whether or not to receive uncertain results and secondary findings. After conducting whole exome sequencing, the findings will be shared with the parent(s). Routine medical care will be provided to patients. The research will study the diagnostic yield of exome sequencing in the prenatal setting for pregnancies with structural anomaly.
Period: Overall Study
Arm/Group | Whole Exome Sequencing
Started | 316
Completed | 316
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregnant Individuals With Fetal Structural Anomalies Were Enrolled, and Followed the Same Procedures: Please note that this is an exploratory study with the outcome of diagnostic yield of exome sequencing in prenatal population and there are no arms. All participants received the same test (exome), and followed the same procedures.
  Whole Exome Sequencing (WES): The Investigators will enroll pregnant women with fetal anomalies detected by ultrasound. Patients will be approached by a maternal-fetal specialist, who has counseled the patient regarding the fetal anomaly that has been detected. Written informed consent will be obtained by the study prenatal genetic counselor. Many patients will have undergone prenatal diagnostic testing in an outside laboratory; in such cases, cells or extracted DNA from the original fetal sample will be used for the purpose of this study. The consent process for prenatal WES will include pre-test counseling and the option of choosing whether or not to receive uncertain results and secondary findings. After conducting whole exome sequencing, the findings will be shared with the parent(s). Routine medical care will be provided to patients. The research will study the diagnostic yield of exome sequencing as a tool for providing genetic information to parents when a prenatal study reveals a fetus with a structural anomaly.
Arm/Group | Pregnant Individuals With Fetal Structural Anomalies Were Enrolled, and Followed the Same Procedures
Number analyzed (Participants) | 316
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 316
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian, Native American, Alaska Native | 0
  Asian | 49
  Black/African American | 3
  Native Hawaiian/Pacific Islander | 0
  White/European American | 115
  Middle Eastern or North African/Mediterranean | 5
  Hispanic/Latino(a) | 49
  More than one race/ethnicity | 25
  Unknown/none of the above | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 316
Number of prenatal patients who consented for a diagnostic exome [Count of Participants; unit: Participants] | 316

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield of Prenatal Exome in Patients With Fetal Structural Anomalies
Description: Number of prenatal patients (pregnancies with a structural anomaly) who got a positive exome result among those who had the exome test. Positive exome result is defined as identification of definitive or probable positive variants which explain prenatal phenotype.
Time Frame: Follow-up was done 6 months after return of exome results.
Population: Pregnant individuals with fetal structural anomalies
Measure: Count of Participants; unit: Participants
Groups:
- Whole Exome Sequencing (WES): Whole Exome Sequencing (WES): The Investigators will enroll pregnant women with fetal anomalies detected by ultrasound. Patients will be approached by a maternal-fetal specialist, who has counseled the patient regarding the fetal anomaly that has been detected. Written informed consent will be obtained by the study prenatal genetic counselor. Many patients will have undergone prenatal diagnostic testing in an outside laboratory; in such cases, cells or extracted DNA from the original fetal sample will be used for the purpose of this study. The consent process for prenatal WES will include pre-test counseling and the option of choosing whether or not to receive uncertain results and secondary findings. After conducting whole exome sequencing, the findings will be shared with the parent(s). Routine medical care will be provided to patients. The research will study diagnostic yield of exome sequencing in prenatal population as a tool for providing genetic information to parents when a prenatal study reveals a fetus with a structural anomaly.
Arm/Group | Whole Exome Sequencing (WES)
Number analyzed (Participants) | 316
Participants | 60

ADVERSE EVENTS:
Time Frame: Data was collected from participants up to 6 months after receiving the results of exome sequencing.
Groups:
- Pregnant Individuals With Fetal Structural Anomalies Were Enrolled, and Followed the Same Procedures: Please note that this is an exploratory study with the outcome of diagnostic yield of exome sequencing in prenatal population and there are no arms. All participants received the same test (exome), and followed the same procedures.
Arm/Group | Pregnant Individuals With Fetal Structural Anomalies Were Enrolled, and Followed the Same Procedures
All-Cause Mortality (participants affected / at risk) | 0/316
Serious Adverse Events (participants affected / at risk) | 0/316
Other Adverse Events (participants affected / at risk) | 0/316

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03482141/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03482141/SAP_001.pdf
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03482141/ICF_003.pdf